CLINICAL TRIAL: NCT00885690
Title: A Multicentre Double-blinded Randomized Head-to-head Study
Brief Title: Comparing the Effects of Sertindole and Olanzapine on Cognition (SEROLA)
Acronym: SEROLA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruitment problems
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg Psychiatric Hospital (Other); Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3.1 - 01-25-09; Eudra CT nr: 2008-008366-13
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic; Cognition
MeSH Terms: conditions — Schizophrenia | interventions — sertindole; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertindole (Active Comparator): Sertindole 16-24 mg
  Interventions: Drug: Sertindole
- Olanzapine (Active Comparator): Olanzapine 10-20 mg
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Sertindole — Sertindole 16-24 mg once daily
  Other Names: Serdolect
  Arms: Sertindole
Drug: Olanzapine — Olanzapine 10-20 mg
  Other Names: Zyprexa
  Arms: Olanzapine

SUMMARY:
Cognition is one of the core symptoms of schizophrenia. This study is a head-to-head trial between olanzapine and sertindole with cognition as primary outcome. The design is a 12-week double-blinded randomized controlled flexible dose study.

ELIGIBILITY:
Inclusion Criteria:

* AnICD-10 schizophrenia diagnosis F20.0-F20.9.
* Contraception.
* A negative pregnancy test for women.
* No known allergy to any of the substances in the study medication
* Baseline QTc < 450 milliseconds for men and < 470 milliseconds for women
* S-potassium and s-magnesium within normal reference range.
* Suboptimally treated on current antipsychotic medication
* Stable dosage of antidepressants and mood stabilizers one month before the inclusion
* Signed informed consent and power of attorney

Exclusion Criteria:

* Withdrawal of consent
* QTc prolongation >500 milliseconds during the study
* Patients with known clinical important cardiovascular disease
* Significant substance abuse
* Earlier partial or non-response in treatment or intolerability to sertindole or olanzapine.
* Calgary Depression Scale score ≥ 7
* Treatment that interferes with the metabolism of sertindole or olanzapine,
* Oxazepam, zopiclone or zolpidem treatment the last 48 hours before cognitive testing
* Prescription of not-allowed medication, or a change in dosage of antidepressant, or mood stabilizers in the study period
* Treatment with an anticholinergic after the first three weeks of the study
* Somatic illness, as judged by investigator, interfering with cognition
* Known risk of narrow angle glaucoma
* Treatment with electroconvulsive therapy (ECT) the last three months before inclusion, or treatment with ECT in the study period
* Treatment with clozapine or depot antipsychotics before inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
CANTAB cognitive test battery | Baseline - 6 and 12 weeks

SECONDARY OUTCOMES:
Fasting glucose, lipid profile, HbA1c, body weight, abdominal circumference, blood pressure | Baseline - 6 and 12 weeks
PANSS, CGI, Sf-36 (quality of life), GAF (social function), UKU (side effects), DAI (attitude towards medicine), Beck's insight scale, Specific Level of Functioning (SLOF) | Baseline, 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: René Nielsen, M.D., Principal Investigator — Aalborg Psychiatric Hospital, Aarhus University Hospital
Locations (2):
- Aalborg Psychiatric Hospital, Aalborg, Denmark
- Universitets Allmänna Sjukhuset, Malmø UMAS, Malmo, Sweden